CLINICAL TRIAL: NCT01764958
Title: Association Between Mother-Infant Attunement During Interaction and the Quality of General Movements and Motor Development of Preterm Infants
Brief Title: Association Between Mother-Infant Attunement During Interaction and the Quality of General Movements
Status: Completed | Type: Observational
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Other Study IDs: sponsor
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2012-04

CONDITIONS: Premature Birth
Keywords: mother-infant interaction; general movements; preterm infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- preterm infants and their mothers: Inclusion criteria are: preterm infants born between 26-34 weeks of gestation, whose mothers speak and write Hebrew fluently. Exclusion criteria are: preterm infants who suffer from perinatal asphyxia, genetic or metabolic diseases, necrotizing colitis that requires operation, intra uterine growth retardation, deafness, retinopathy of prematurity (ROP) or major congenital defects.
  Infants and their mothers will be recruited from child developmental centers and Pediatric Clinics of Maccabi. No intervention is included in the research.

SUMMARY:
The proposed research has the potential of contributing to the limited empirical literature on the relationship between maternal sensitivity and motor development of preterm infants. If indeed maternal attuned behaviors will be found to be associated with the quality of motor development, such a finding will support the effectiveness of physical therapy in guiding caregivers to attune their holding and touch of preterm infants.

We hypothesize that mothers and infants' attunement during observed interaction will be related to the quality of preterm infants' spontaneous movements in the following ways: First, better maternal attunement to the infants needs, and in particular attunement of holding and touch will be associated with better quality of spontaneous movements of the infants. Second, more initiations and/or involvement of infants in interaction will be associated with better maternal attunement to the infant. Third, more initiations and/or involvement of infants in interaction will be associated with better quality of spontaneous movements and better achievements in developmental milestone. All hypotheses will be examined while controlling for maternal use of SSC method during hospitalization after birth and family demographic backgrounds.

DETAILED DESCRIPTION:
Sixty preterm infants at 3-4 months of corrected age and their mothers will be recruited. Infants will be evaluated for their spontaneous movements and their developmental milestones achievement, and mothers and infants will be evaluated for their attunement during observed interaction, especially on maternal attunement in holding and touching their infants. Mothers will report on demographic background of the family, temperament of their infants and previous Skin to Skin Contact treatment in the Neonatal Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:preterm infants born between 26-34 weeks of gestation, whose mothers speak and write Hebrew fluently.

-

Exclusion Criteria:preterm infants who suffer from perinatal asphyxia, genetic or metabolic diseases, necrotizing colitis that requires operation, intra uterine growth retardation, deafness, retinopathy of prematurity (ROP) or major congenital defects.

-

Ages: 4 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants at a corrected age of 3-4 months and their mothers
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Better maternal attunement of holding and touch will be associated with better quality of spontaneous movements of the infants. | Assesed at 3-4 months corrected age of the infants
  Infants are videotapes for General Movements Mothers and infants are videotapes for 10 minutes of free interaction

SECONDARY OUTCOMES:
More initiations and/or involvement of infants during the interaction will be associated with better quality of spontaneous movements of the infants and better achievement in developmental milestones. | 3-4 months corrected age of the infants
  in addition to General Movements and Interaction, developmental milestones will be assessed using the Alberta Infant Motor development Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Orna Lev enacab, BPT, Principal Investigator — Assuta Hospital, Tel Aviv
Locations (1):
- Maccabi Healthcare services, Naẕerat ‘Illit, Israel